CLINICAL TRIAL: NCT00448981
Title: Stopping URIs and Flu in the Family: The Stuffy Trial
Brief Title: Stopping Upper Respiratory Infections and Flu in the Family: The Stuffy Trial
Acronym: STUFFY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCEZID-5033; 1U01CI000442-01 (NIH)
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Respiratory Tract Infections; Common Cold
Keywords: Preventing upper respiratory tract infections; Preventing influenza; Preventing the common cold; Hand hygiene and upper respiratory infections; Mask use in preventing upper respiratory infections
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold | interventions — Hand Hygiene; Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Hand hygiene and educational material
Device: Mask, alcohol and hand sanitizer

SUMMARY:
Colds and flu cause much loss of work and school. The purpose of this study is to try to reduce the transmission of colds and flu among household members with one of three interventions: some educational material, educational material and use of alcohol hand sanitizers, and educational material and use of alcohol hand sanitizers as well as face masks when somebody has symptoms of the flu. We will recruit 450 households in Northern Manhattan and each household will be randomly assigned to one of these three groups. We will then follow these households for 15 months to see how often they get cold and flu symptoms. We will also look at antibiotic use practices for symptoms of colds and influenza ; household member knowledge of prevention and treatment strategies for pandemic influenza and viral URIs; and rates of influenza vaccination among household members. When someone in the study has serious flu symptoms such as a high fever and cough or sore throat, we will also obtain a nasal culture (by swabbing the nose) to see if there is flu virus present.

DETAILED DESCRIPTION:
Although 'colds' and seasonal influenza are clinically very different diseases from pandemic influenza, they share common transmission pathways and the community level interventions needed to reduce both seasonal flu, common viral upper respiratory infections and pandemic influenza are likely to be similar.

Aims of this project are to compare the impact of two household level interventions (an alcohol based hand sanitizer with or without face masks) on six outcomes: incidence and strains of virologically confirmed influenza in study households; rates of symptoms; number of secondary cases in households; antibiotic use practices for symptoms of influenza and other viral upper respiratory infections; household member knowledge of prevention and treatment strategies for pandemic influenza and viral upper respiratory infections; and rates of influenza vaccination among household members.

450 households in northern Manhattan (primarily recently immigrated Hispanics) will be randomized to three groups: control (receiving only a pamphlet on influenza prevention), alcohol hand sanitizer, and sanitizer plus face masks. Symptoms of influenza will be monitored daily for 15 months using ecological momentary assessment technology. Virologic cultures will be obtained from persons with flu symptoms (fever >100 degrees F., sore throat and/or cough). Antibiotic use practices, knowledge, and vaccination rates will be assessed by survey using piloted, psychometrically sound instruments. For this cluster randomization design with randomized intervention on the household level, outcomes will be measured at the individual and household level using generalized linear mixed model for counts response with a Poisson distribution and other appropriate multivariate techniques to control for confounding.

Comparison(s): The purpose of this study is to try to reduce the transmission of colds and flu among household members with one of three interventions: comparison of transmission in groups receiving educational material only to a group receiving educational material and instructed to use alcohol hand sanitizers to a group receiving educational material and instructed to use alcohol hand sanitizers as well as face masks when somebody has symptoms of the flu

ELIGIBILITY:
Inclusion Criteria:

* Households which include at least three persons, at least one of whom is a preschool child, living in Northern Manhattan, have a telephone, speak Spanish or English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2788 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Rates of virologically confirmed influenza and influenza vaccination
Rates of influenza-like symptoms
Knowledge and attitudes about influenza and the common cold and antibiotic use practices.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Larson, RN,PhD, Principal Investigator — Columbia University School of Nursing
Locations (1):
- Columbia University School of Nursing, New York, New York, United States

REFERENCES:
- [Derived] Cohen B, Ferng YH, Wong-McLoughlin J, Jia H, Morse SS, Larson EL. Predictors of flu vaccination among urban Hispanic children and adults. J Epidemiol Community Health. 2012 Mar;66(3):204-9. doi: 10.1136/jech.2009.099879. Epub 2010 Sep 29. PMID 20881023